CLINICAL TRIAL: NCT05919914
Title: The Immediate Effects of a Wrist Extensors Exercise With Blood Flow Restriction BFR in Lateral Elbow Tendinopathy. A Randomized Controlled Trial.
Brief Title: The Effects of a Wrist Extensors Exercise With Blood Flow Restriction (BFR) in Lateral Elbow Tendinopathy.
Acronym: BFR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of West Attica (Other)
Responsible Party: Principal Investigator, Stefanos Karanasios, Principal Investigator, University of West Attica
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 11168 - 06/02/2023
Record Dates: First submitted 2023-06-12; First posted 2023-06-26 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Lateral Epicondylitis
Keywords: tennis elbow; pain threshold; elbow tendinopathy; BFR; hypoalgesia
MeSH Terms: conditions — Tennis Elbow; Elbow Tendinopathy | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wrist extensor exercise with Blood Flow Restriction (Experimental): Blood flow restriction training. Patients will execute a wrist extension exercise on standing position with the elbow extended. The load (dumbbells) will be set according to a pain monitoring approach ( exercise should not provoke pain >2/10) during wrist extension. Load is increased by 0.5 to 1kg. We will allow a 30 sec break. The session starts by calculating the arterial occlusion pressure in the standard anatomical position. Participants rest in the standing position for 3-5 minutes before measurement to ensure restoration of blood flow circulation and a cuff is placed in the most proximal part of their dominant upper-limb. BFR application is conducted by using an automatic personalized tourniquet system (Mad-Up Pro, France).
  An 40% occlusion pressure is set and subjects perform 4 sets of wrist extension (30-15-15-15 reps).
  Interventions: Other: Exercise with Blood Flow Restriction (BFR)
- Wrist extensor exercise without Blood Flow Restriction (Active Comparator): Patients will execute a wrist extension exercise on standing position with the elbow extended. The load (dumbbells) will be set according to a pain monitoring approach ( exercise should not provoke pain >2/10) during wrist extension. Load is increased by 0.5 to 1kg. We will allow a 30 sec break.
  Interventions: Other: Exercise without Blood Flow Restriction (BFR)

INTERVENTIONS:
Other: Exercise with Blood Flow Restriction (BFR) — Wrist extensor exercise (concentric - eccentric) with BFR. BFR involves the reduction of blood flow to working skeletal muscle by applying a flexible cuff to the most proximal portions of a person's arms or legs that results in decreased arterial flow to the exercising muscle and occluded venous return back to the central circulation.
  Arms: Wrist extensor exercise with Blood Flow Restriction
Other: Exercise without Blood Flow Restriction (BFR) — Wrist extensor exercise (concentric - eccentric)
  Arms: Wrist extensor exercise without Blood Flow Restriction

SUMMARY:
A randomized cross-over trial comparing the immediate effects of a wrist extensor exercise with and without blood flow restriction (BFR) on pain perception in patients with lateral elbow tendinopathy (LET).

DETAILED DESCRIPTION:
Patients with LET will participate in the study performing an exercise with and without blood flow restriction (BFR) in a randomized order (two occasions). A target of 20 patients for enrollment has been set for 80% power, p<0.05 (Effect size= 1). Two interventions will be used lasting 40 minutes each.

Intervention: A wrist extension exercise (concentric-eccentric) with Blood Flow Restriction (30-15-15-15 reps). Exercises will be performed using dumbbells according to a pain monitoring approach (<2/10 in numerical pain rating scale).

Control Group: A wrist extension exercise (concentric-eccentric) without Blood Flow Restriction (30-15-15-15 reps). Exercises will be performed using dumbbells according to a pain monitoring approach (<2/10 in numerical pain rating scale).

Primary outcomes: pressure pain thresholds lateral epicondyle, cervical spine and tibialis anterior (bilateral).

Secondary outcome: pain free grip strength

ELIGIBILITY:
Inclusion Criteria:

* Men and women diagnosed with Lateral Elbow Tendinopathy (LET)
* Symptoms for over 2 weeks
* Pain provoked by palpation on the lateral epicondyle
* Positive: Cohen's test, Maudsley test, Mill's test
* decrease in pain grip strength >5% in elbow extension compared to flexion

Exclusion Criteria:

* Shoulder tendinopathy
* Cervical radiculopathy
* Rheumatoid arthritis
* Neurological deficit
* Radial nerve entrapment
* Past treatment for the elbow before entering the study
* Professional athletes
* Lateral elbow tendinopathy of the same side in the last 3 years
* Serious cardiovascular diseases
* Venous deficiency
* History of heart surgery
* Cancer history
* Breast surgery
* Orthopaedic surgeries during the last 6 months
* Thrombosis
* Body mass Index ≥ 30
* Crohn syndrome
* Family or personal history of pulmonary embolism

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-29 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Pressure pain threshold | Baseline and 30 minutes
  Changes between pre- and post- intervention in Pressure Pain Threshold will be measured using bilateral sites on lateral epicondyle, cervical spine and tibialis anterior. The COMPACT DIGITAL ALGOMETER CAPACITIES TO: 100 lbf / 50 kgf / 500 N, will be used by an independent assessor. The assessor will be blinded to participants' group.

SECONDARY OUTCOMES:
Pain free grip strength (PFGS) | Baseline and 30 minutes
  'Jamar' hand dynamometer was used, calculating the mean value (kilograms) of 3 efforts, separated by 30-second rest intervals with participants lying in supine position and the elbow fully extended

CONTACTS AND LOCATIONS:
Overall Officials: George Gioftsos, PhD, Study Chair — Physiotherapy Department
Locations (1):
- University of West Attica, Aigáleo, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karanasios S, Korakakis V, Moutzouri M, Xergia SA, Tsepis E, Gioftsos G. Low-Load Resistance Training With Blood Flow Restriction Is Effective for Managing Lateral Elbow Tendinopathy: A Randomized, Sham-Controlled Trial. J Orthop Sports Phys Ther. 2022 Dec;52(12):803-825. doi: 10.2519/jospt.2022.11211. Epub 2022 Sep 13. PMID 36099170
- [Background] Karanasios S, Lignos I, Gioftsos G. Wrist Extensor Training With Blood Flow Restriction for the Management of Lateral Elbow Tendinopathy: A Case Report. Cureus. 2023 Feb 25;15(2):e35468. doi: 10.7759/cureus.35468. eCollection 2023 Feb. PMID 36999107
- [Background] Peterson M, Butler S, Eriksson M, Svardsudd K. A randomized controlled trial of eccentric vs. concentric graded exercise in chronic tennis elbow (lateral elbow tendinopathy). Clin Rehabil. 2014 Sep;28(9):862-72. doi: 10.1177/0269215514527595. Epub 2014 Mar 14. PMID 24634444
- [Background] Yoon SY, Kim YW, Shin IS, Kang S, Moon HI, Lee SC. The Beneficial Effects of Eccentric Exercise in the Management of Lateral Elbow Tendinopathy: A Systematic Review and Meta-Analysis. J Clin Med. 2021 Sep 1;10(17):3968. doi: 10.3390/jcm10173968. PMID 34501416
- [Background] Bisset L, Coombes B, Vicenzino B. Tennis elbow. BMJ Clin Evid. 2011 Jun 27;2011:1117. PMID 21708051
- [Background] Lee JH, Kim TH, Lim KB. Effects of eccentric control exercise for wrist extensor and shoulder stabilization exercise on the pain and functions of tennis elbow. J Phys Ther Sci. 2018 Apr;30(4):590-594. doi: 10.1589/jpts.30.590. Epub 2018 Apr 20. PMID 29706713
- [Background] Coombes BK, Bisset L, Vicenzino B. Management of Lateral Elbow Tendinopathy: One Size Does Not Fit All. J Orthop Sports Phys Ther. 2015 Nov;45(11):938-49. doi: 10.2519/jospt.2015.5841. Epub 2015 Sep 17. PMID 26381484